CLINICAL TRIAL: NCT04593654
Title: Dosing of Thromboprophylaxis and Mortality in Critically Ill COVID-19 Patients - More Patients Included and 90-day Follow up
Brief Title: Dosing of Thromboprophylaxis and Mortality in Critically Ill COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sandra Jonmarker, Principal investigator, MD, PhD-student, Karolinska Institutet
Other Study IDs: Thromboprophylaxis COVID-19
Record Dates: First submitted 2020-10-16; First posted 2020-10-20 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Covid19; Thromboembolism
Keywords: Pulmonary embolism; Anticoagulation; Critical Care; Bleeding; Ischemic stroke
MeSH Terms: conditions — COVID-19; Thromboembolism; Pulmonary Embolism; Hemorrhage; Ischemic Stroke | interventions — Dalteparin; Tinzaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low dose thromboprophylaxis: Daily dose of 2500-4500 IU tinzaparin or 2500-5000 IU dalteparin
  Interventions: Drug: Dose of tinzaparin or dalteparin
- medium dose thromboprophylaxis: Daily dose of >4500 IU but <175 IU/kg of body weight tinzaparin or >5000 IU but <200 IU/kg of body weight dalteparin
  Interventions: Drug: Dose of tinzaparin or dalteparin
- high dose thromboprophylaxis: Daily dose of ≥ 175 IU/kg of body weight tinzaparin or ≥200 IU/kg of body weight dalteparin
  Interventions: Drug: Dose of tinzaparin or dalteparin

INTERVENTIONS:
Drug: Dose of tinzaparin or dalteparin — The patients will be categorised into three groups depending on initial dose of thromboprophylaxis in the ICU
  Other Names: Innohep/Fragmin

SUMMARY:
The aim of the study is to associate dose of thromboprophylaxis with outcome in critically ill COVID-19 patients. This will be done by associating dose of thromboprophylaxis with 28-day mortality, survival outside ICU, thromboembolic event and bleeding complications.This was done in our earlier study for patients admitted in March and April (Clinicaltrials.gov NCT04412304 June 2 2020) but now we will include the patients admitted in May, June and half of July and we will ad the outcome of 90-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* laboratory confirmed positive test for SARS-CoV-2
* admitted to ICU because of respiratory failure caused by Covid-19

Exclusion Criteria:

* patients with treatment for thromboembolic complications at arrival to the ICU
* short ICU length of stay defined as discharged the same date as ICU admission
* patients without initial thromboprophylaxis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort study of the critically ill Covid-19 patients admitted to ICU at Södersjukhuset, Stockholm from1st of March to 15 of July
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days from ICU-admission
  28-day mortality from admission to ICU. Discontinue of ICU-care to palliative care counts as death.

SECONDARY OUTCOMES:
Incidence of thromboembolic events | 28 days from ICU-admission
  Thromboembolic events are defined as pulmonary emboli (PE), deep venous thrombus (DVT) and ischemic stroke. PE is defined as PE verified by computer tomography or by findings of acute strain of the right heart on echocardiography combined with a clinical interpretation of the patients deteriorating as a probable PE stated in the medical records. DVT is defined as DVT verified with ultrasound. Ischemic stroke is defined as ischemic stroke verified by computer tomography.
Incidence of bleeding events | 28 days from ICU-admission
  The event of bleeding will be defined by WHO modified bleeding scale as 1-4
ICU-free days alive from ICU-admission | 28 days from ICU-admission
  ICU-free days alive during 28 days from ICU-admission. Counts as 0 days if discharged to ward for palliative treatment.
90-day mortality | 90 days from ICU-admission
  90-day mortality from admission to ICU.

OTHER OUTCOMES:
Fibrin-D-dimer levels | 28 days from ICU-admission
  Median value of Fibrin-D-dimer

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jonmarker, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Södersjukhuset, Stockholm, Sweden

REFERENCES:
- [Derived] Jonmarker S, Litorell J, Dahlberg M, Stackelberg O, Everhov AH, Soderberg M, Rubenson-Wahlin R, Gunther M, Martensson J, Hollenberg J, Joelsson-Alm E, Cronhjort M. An observational study of intermediate- or high-dose thromboprophylaxis for critically ill COVID-19 patients. Acta Anaesthesiol Scand. 2022 Mar;66(3):365-374. doi: 10.1111/aas.14013. Epub 2021 Dec 16. PMID 34875111